CLINICAL TRIAL: NCT06251791
Title: Exploring The Impact Of Inspiratory Muscle Training on Expiratory Muscle Thickness During Intensive Care Patients
Brief Title: Inspiratory Muscle Training and Expiratory Muscle Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Reyhan Kaygusuz, Principal Investigator, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IMT on abdominal muscle
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Intensive Care Unit Syndrome; Muscle Weakness; Rehabilitation
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Parallel Assignment Randomized Healthy participants
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental (Experimental): Experimental: Conventional Physiotherapy In the intensive care unit and who had mechanical ventilation for more than 48 hours and who were extubated. In this group addition to conventional physiotherapy inspiratory muscle training will be performed with the threshold-loaded inspiratory muscle training device, starting at 30% of the maximum inspiratory mouth pressure value, during 5 days, in 2 sessions, 4 sets per day, 6-8 breaths in each set and 2 minutes of rest between sets.
  Interventions: Other: conventional physiotherapy+ IMT
- Conventional (Experimental): In this group will apply only conventional physiotherapy. Conventional physiotherapy to contain breathing and,thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization. Conventional physiotherapy apply for 5 days after extubation period 1 time a day.
  Interventions: Other: conventional physiotherapy
- Healthy controls (No Intervention): There is no intervention in this group. Baseline measurements are to compare with experimental groups.

INTERVENTIONS:
Other: conventional physiotherapy+ IMT — Conventional Physiotherapy to contain breathing and thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization in 1 time a day. Conventional Physiotherapy to contain breathing and thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization in 1 time a day. In this group addition to conventional physiotherapy inspiratory muscle training will be performed with the threshold-loaded inspiratory muscle training device, starting at 30% of the maximum inspiratory mouth pressure value, during 5 days, in 2 sessions, 4 sets per day, 6-8 breaths in each set and 2 minutes of rest between sets.
  Arms: Experimental
Other: conventional physiotherapy — Conventional Physiotherapy to contain breathing and thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization in 1 time a day. Conventional Physiotherapy to contain breathing and thoracal expansion exercises, bronchial hygiene techniques and gradual mobilization in 1 time a day.
  Arms: Conventional

SUMMARY:
the specific effect of IMT on expiratory muscle strength and abdominal wall thickness during weaning remains unclear. To address this significant research gap, the primary objective of our study was to evaluate the effect of IMT after extubation on expiratory muscle strength and abdominal muscle thickness in respiratory ICU patients. On the other hand the investigators established reference values for ultrasonographic measurements in healthy control subjects as a comparative arm. To the best of our knowledge, this is the first study to examine the ultrasonographic effects of IMT on the expiratory muscle thickness after extubation. The investigators believe that our study may contribute to related literature in this context and guide future research as a pioneer with its unique value.

DETAILED DESCRIPTION:
the specific effect of IMT on expiratory muscle strength and abdominal wall thickness during weaning remains unclear. To address this significant research gap, the primary objective of our study was to evaluate the effect of IMT after extubation on expiratory muscle strength and abdominal muscle thickness in respiratory ICU patients. On the other hand the investigators established reference values for ultrasonographic measurements in healthy control subjects as a comparative arm. To the best of our knowledge, this is the first study to examine the ultrasonographic effects of IMT on the expiratory muscle thickness after extubation. The investigators believe that our study may contribute to related literature in this context and guide future research as a pioneer with its unique value. In this single-blind randomized controlled study, 20 patients were divided into two groups: IMT and conventional physiotherapy(CP). In order to establish normative data for abdominal muscle thickness, ten healthy controls were included in the study. The CP group received CP and the IMT group received CP+IMT for five days following extubation. The thicknesses of the external oblique abdominal(EOA),internal oblique sbdominal(IOA), transversus abdominus (TRA) and rectus abdominis (RA) muscleswere evaluated The maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) were recorded.

ELIGIBILITY:
Inclusion Criteria:

* For Patients Group Inclusion Criteria:

  * Needing mechanical ventilation support longer than 2 days,
  * Alert and Riker Sedation Agitation Score >4
  * Being hemodynamically stable (HR<140 beats/min, BP stable)
  * Dobutamine and minimal vasopressor use
  * Fever of 36.5-38.5
  * Body Mass Index <40 m2/cm,
  * FiO2 of 0.5 or less,
  * Absence of myocardial ischemia.

Exclusion Criteria:

* For Patients Group Exclusion Criteria:

  * Noncooperation
  * Phrenic nerve damage
  * Chest wall trauma and/or deformity to prevent diaphragmatic movement
  * Progressive neuromuscular disease with respiratory involvement
  * There is enough secretion to require more than one aspiration every hour.
  * Patients using sedative drugs continuously
  * High-dose cortisol use
  * Using a home mechanical ventilator before mechanical ventilation in intensive care unit

For Healthy Group Inclusion Criteria:

* With the control and intervention group, age, characteristics and characteristics,
* Chronic system and no ongoing treatment,
* Body mass index not 40 kg/m2,
* 18-80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Abdominal Muscle Thickness | Change from baseline Maximal inspiratory and expiratory pressure at 5th day]
  Eksternal Oblique, Internal Oblique, Transverses Abdominus and rectus abdominus Ultrasonografic mesasurements

SECONDARY OUTCOMES:
Maximal inspiratory and expiratory pressure | Change from baseline Maximal inspiratory and expiratory pressure at 5th day]
  Intraoral pressures measured at maximal respiration against a valve that closes the airway during maximal inspiration pressure and expiration. Maximal inspiration pressure is the highest pressure created to open closed alveoli at the residual volume level. In our study, respiratory muscle strength will be performed using a portable, electronic mouth pressure measuring with device. For the test, the applied person is given maximum expiration and at the end of this, the airway is closed with a valve and the person is asked to make maximum inspiration and continue it for 1-3 seconds. In the maximal expiration pressure measurement, after maximal inspiration, the person is asked to make a maximal expiration for 1-3 seconds against the closed airway. The best of the three measurements is selected. There should be no more than 10% or more than 10 cmH2O difference between the two best measured

CONTACTS AND LOCATIONS:
Overall Officials: barış yılmaz, MD, Study Chair — Sureyyapasa Chest Diseases and Thoracic Surgery Training and Research Hospital
Locations (1):
- Istanbul Demiroglu University, Istanbul, Şişli, Turkey (Türkiye)